CLINICAL TRIAL: NCT02993367
Title: The Efficacy of Butylphthalide Soft Capsules in Patents With VCIND:A Randomized, Double-blind,and Neuroimaging Study
Brief Title: The Efficacy of Butylphthalide Soft Capsules in Patents With VCIND
Acronym: EBSCPVCIND
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yifei Zhu, Clinical Professor, The Second Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZYF55688
Record Dates: First submitted 2016-12-08; First posted 2016-12-15 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Vascular Cognitive Impairment no Dementia
Keywords: Butylphthalide Soft Capsules; VCIND; fMRI

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the Butylphthalide Soft Capsules group (Experimental): 600mg Butylphthalide Soft Capsules/day,po tid,period of 6 months
  Interventions: Drug: Butylphthalide Soft Capsules
- the placebo group (Placebo Comparator): 60mg Butylphthalide Soft Capsules/day,po tid,period of 6 months
  Interventions: Drug: Placebo Butylphthalide Soft Capsules

INTERVENTIONS:
Drug: Butylphthalide Soft Capsules — DL-3-n-butylphthalide (NBP) (Fig. 1) is a synthetic chiral compound containing L- and D-isomers of butylphthalide.Butylphthalide Soft Capsules is the oral preparation.
  Arms: the Butylphthalide Soft Capsules group
Drug: Placebo Butylphthalide Soft Capsules
  Arms: the placebo group

SUMMARY:
Vascular cognitive impairment no dementia (VCIND) is very common among the aged and tends to progress to dementia, but there have been no proper large-scale intervention trials dedicated to it. VCIND caused by subcortical ischemic small vessel disease (hereinafter, subcortical VCIND) represents a relatively homogeneous disease process and is a suitable target for therapeutic trials investigating VCIND. Preclinical trials showed that Butylphthalide Soft Capsules is effective for cognitive impairment of vascular origin. In this randomized, double-blind, placebo-controlled trial, the investigators apply fMRI study the effects of Butylphthalide Soft Capsules in patients with VCIND.

ELIGIBILITY:
Inclusion Criteria:

* Literate Han Chinese aged from 40 to 65 years
* MMSE ≥24
* Normal or slightly impaired activities of daily living
* The MRI entry criteria are as follows:

  * Subcortical small infarcts (3-20 mm in diameter),or one or more strategically located subcortical small infarcts in the caudate nucleus globus pallidus, or thalamus
  * Absence of cortical and watershed infarcts, hemorrhages, hydrocephalus, and WMLs with specific causes (e.g., multiple sclerosis); and
  * No hippocampal or entorhinal cortex atrophy (scored 0 according to medial temporal lobe atrophy scale of Scheltens)

Exclusion Criteria:

* Patients with Diabetes mellitus
* Disorders other than subcortical VCIND that may affect cognition; the score of Hamilton depression scale more than 17 or schizophrenia
* Clinically significant gastrointestinal, renal, hepatic, respiratory, infectious, endocrine, or cardiovascular system disease; cancer; alcoholism; drug addiction; use of medications that may affect cognitive functioning
* Known hypersensitivity to celery
* Inability to undergo a brain MRI

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
change of Cognitive function | Time points 0, 1, 3 and 6 months

SECONDARY OUTCOMES:
change of brain function | Time point at 0, 1, 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yifei Zhu, M.D., Principal Investigator — The Second Hospital of Hebei Medical University
Locations (1):
- Second Affiliated Hospital of Hebei medical university, Shijiazhuang, Hebei, China

REFERENCES:
- [Result] Jia J, Wei C, Liang J, Zhou A, Zuo X, Song H, Wu L, Chen X, Chen S, Zhang J, Wu J, Wang K, Chu L, Peng D, Lv P, Guo H, Niu X, Chen Y, Dong W, Han X, Fang B, Peng M, Li D, Jia Q, Huang L. The effects of DL-3-n-butylphthalide in patients with vascular cognitive impairment without dementia caused by subcortical ischemic small vessel disease: A multicentre, randomized, double-blind, placebo-controlled trial. Alzheimers Dement. 2016 Feb;12(2):89-99. doi: 10.1016/j.jalz.2015.04.010. Epub 2015 Jun 15. PMID 26086183